CLINICAL TRIAL: NCT03986333
Title: Validity, Reliability and Responsiveness to Change of the French Version of the Drooling Impact Scale in a Pediatric Cerebral Palsy Population.
Brief Title: Validation of the French Version of the Drooling Impact Scale in a Pediatric Cerebral Palsy Population
Status: Completed | Type: Observational
Sponsor: Centre Médico-Chirurgical de Réadaptation des Massues Croix Rouge Française (Other)
Responsible Party: Sponsor
Other Study IDs: DROOLING
Record Dates: First submitted 2019-05-13; First posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-05

CONDITIONS: Cerebral Palsy; Drooling
MeSH Terms: conditions — Cerebral Palsy; Sialorrhea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Children whose drooling was expected to remain relatively stable over 1 month
- Intervention: Children receiving a treatment to reduce their drooling

SUMMARY:
The aim of this study is to present the French translation of the Drooling Impact Scale (DIS-F) and to explore its validity, reliability and responsiveness to change in a group of children with Cerebral Palsy (CP)

DETAILED DESCRIPTION:
Drooling in children with CP is likely underestimated and under treated. It is an over-handicap for these children, because it causes many complications and may lead to a decline in self-esteem and to social isolation, altering the quality of life for patients and families. The therapeutic arsenal for the management of drooling includes rehabilitation techniques, oral drug treatments, local treatments or surgical treatments whose effectiveness is variable. In order to evaluate the efficacy of these therapies, standardized and valid assessment tools must be used. The Drooling Impact Scale (DIS) developed by Dr. Sue Reid's team in Melbourne in 2008, shows good validity and sensitivity to change, especially after botulinum toxin injection. It is commonly used in English-speaking studies, but no validation in French is available yet.

The aim of this study is to present the French translation of the Drooling Impact Scale (DIS-F) and to explore its validity, reliability and responsiveness to change in a group of children with CP.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral palsy
* Hypersialorrhea
* No change in content and frequency of speech therapy for three months following baseline
* At least 1 out of 2 parents must have a clear understanding of french language
* Oral consent

Exclusion Criteria:

* No clear understanding of french language

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Fifty-five children were included, 33 in the stable group and 22 in the intervention group.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in Drooling Impact Scale | Control group : baseline and 1 month later. Intervention group : baseline and 1 month after treatment
  The severity of drooling is assessed from the parents perception, by the Drooling Impact Scale. This scale consists of a set of ten items exploring the impact of drooling on daily life activities and relationships, each measured on a scale of 1 to 10 (1 representing the lowest impact of drooling, 10 the highest).

SECONDARY OUTCOMES:
Internal consistency | All groups : at inclusion
  Internal consistency was assessed by calculating the Cronbach's alpha coefficient from scores obtained at inclusion. A correlation coefficient of at least 0.7 was defined as indicative of adequate inter-relatedness of items. The Pearson correlation matrix was used to define the linear relationships between items.
Test-retest reliability | Control group : baseline and 1 month later
  The Lin concordance correlation coefficient was used to compute the level of agreement between the two assessments. In addition, the Bland-Altman limits-of-agreement method for assessing test-retest reliability was used as a complementary approach.
Responsiveness to change | Intervention group : baseline and 1 month after treatment.
  An estimate of the responsiveness or sensitivity to change of the measure was obtained using four statistical methods : effect size, standardized response mean,Guyatt responsiveness statistics, unpaired t-test (Wilcoxon test).

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle Chaléat-Valayer, PhD, Principal Investigator — CMCR des Massues Croix rouge française
Locations (6):
- France (6):
  - Centre d'Education Motrice Jean-Marie Arnion - Odynéo, Dommartin
  - Centre d'Education Motrice Henry Gormand, Écully
  - Centre Hospitalier Universitaire Hôpital Nord, La Tronche
  - Croix rouge française Centre Médico-Chirurgical de Réadaptation des Massues, Lyon
  - AP-HM Hôpital de la Timone, Marseille
  - Centre Hospitalier Universitaire de Nîmes, Nîmes